CLINICAL TRIAL: NCT01514448
Title: An Open Label, Single Arm Trial to Evaluate Patients With Metastatic Renal Cell Carcinoma Treated With Everolimus After Failure of First Line Therapy With Sunitinib or Pazopanib
Brief Title: Safety and Efficacy of Everolimus in Metastatic Renal Cell Carcinoma After Failure of First Line Therapy With Sunitinib or Pazopanib
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001LDE43; 2011-003416-23 (EudraCT Number)
Record Dates: First submitted 2012-01-17; First posted 2012-01-23 (Estimated); Results first posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Metastatic Renal Cell Carcinoma (mRCC)
Keywords: Kidney cancer; mRCC; metastic renal cell carcinoma; everolimus; sunitinib; pazopanib
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Everolimus (Experimental): Everolimus 10 mg orally once daily until disease progression, occurrence of intolerable toxicity, start of another anticancer treatment or withdrawn consent.
  Interventions: Drug: Everolimus (RAD001)

INTERVENTIONS:
Drug: Everolimus (RAD001) — Everolimus was used as commercially available formulated tablets of 10 mg strength
  Other Names: RAD001

SUMMARY:
Patients with metastatic renal cell carcinoma (mRCC) who failed first-line therapy with sunitinib or pazopanib was treated with everolimus. Efficacy and safety of everolimus was evaluated in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced renal cell carcinoma of a histological or cytological confirmation of clear cell renal carcinoma.
* Progression during or after a treatment with sunitinib or pazopanib given in a 1st line treatment situation for mRCC.
* Patients scheduled for treatment with everolimus.
* Patients with at least one measurable lesion at baseline as per RECIST v1.1.

Exclusion Criteria:

* Patients who have received >1 prior systemic treatment for their metastatic RCC. Prior systemic treatment in an adjuvant setting is allowed.
* Patients who have previously received systemic mTOR inhibitors (e.g. sirolimus, temsirolimus, everolimus).
* Patients who are using other investigational agents or who had received investigational drugs ≤ 2 weeks prior to study treatment start.
* Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-05-21 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2016-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Germany (13):
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Hof
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Langen
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Ravensburg
  - Novartis Investigative Site, Velbert
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Wolfsburg

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Single arm study of everolimus broken down into 2 subgroups for analyses and safety based on failed 1st line therapy (sunitinib or pazopanib) prior to starting study.
Groups:
- 1st Line SUN: Patients that failed 1st line therapy Sunitinib (SUN) prior to starting study. Patients were on Everolimus 10 mg orally once daily until disease progression, occurrence of intolerable toxicity, start of another anticancer treatment or withdrawn consent.
- 1st Line PAZ: Patients that failed 1st line therapy Pazopanib (PAZ) prior to starting study. Patients were on Everolimus 10 mg orally once daily until disease progression, occurrence of intolerable toxicity, start of another anticancer treatment or withdrawn consent.
Period: Overall Study
Arm/Group | 1st Line SUN | 1st Line PAZ
Started | 16 | 13
Full Analysis Set (FAS) | 12 | 13
Completed | 4 | 5
Not Completed | 12 | 8
Not completed — Death | 7 | 8
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — New Cancer Therapy | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographic and other baseline data (including disease characteristics) were summarized descriptively for all patients for the FAS. The full analysis set (FAS) consisted of all patients who received at least one dose of everolimus.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1st Line SUN | 1st Line PAZ | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (6.3) | 71.3 (6.0) | 69.2 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 6 | 11 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Progression-free Patients by Month 6
Description: Percentage of progression-free patients by month 6 after starting everolimus treatment. For the purpose of the binomial design of the study, a patient being 'progression-free' will be defined as a patient without disease progression by month 6 whereas a subject with progressive disease by month 6 will not be counted as 'progression-free'. The primary variable was derived from radiologic tumor assessments according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1.) Disease progression was either 1) a 20% increase in the sum of the longest diameter of all target lesions, taking as reference the smallest sum of the longest diameters of all target lesions recorded at or after baseline (minimum absolute increase 5 mm in sum) or 2) the appearance of a new lesion or 3) the unequivocal progression of non-target lesions overall.
Time Frame: Month 6
Population: Full Analysis Set (FAS) consisted of all patients who received at least one dose of everolimus.
Measure: Number; unit: Percentage of participants
Arm/Group | 1st Line SUN | 1st Line PAZ
Number analyzed (Participants) | 12 | 13
Percentage of participants | 8.3 | 46.2

2. Secondary Outcome: Percentage of Patients With Overall Response Rate (ORR) Treated With Everolimus After Failure of First-line Sunitinib or Pazopanib Therapy at Month 6
Description: Overall response rate (ORR) is the Percentage of patients with a best overall response of complete response (CR) or partial response (PR) by month 6. ORR was assessed according to RECIST 1.1 criteria. Partial response (PR) required at least a 30% decrease in the sum of the longest diameters of all target lesions, taking as reference the baseline sum of the longest diameters. Complete response (CR) required a disappearance of all target and non-target lesions.
Time Frame: Month 6
Population: Full Analysis Set (FAS) consisted of all patients who received at least one dose of everolimus.
Measure: Number; unit: percentage of participants
Arm/Group | 1st Line SUN | 1st Line PAZ
Number analyzed (Participants) | 12 | 13
percentage of participants | 0.0 | 0.0

3. Secondary Outcome: Progression-Free Survival (PFS) as the Time Interval Between First Intake of Everolimus and First Documented Disease Progression or Death Due to Any Cause at 24 Months
Description: Progression-free survival (PFS) is the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause. If a patient did not have an event, progression-free survival was censored at the date of last adequate tumor assessment
Time Frame: 24 months
Population: Full Analysis Set (FAS) consisted of all patients who received at least one dose of everolimus.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | 1st Line SUN | 1st Line PAZ
Number analyzed (Participants) | 12 | 13
months | 2.8 [2.6 to 3.1] | 8.0 [3.0 to 10.3]

4. Secondary Outcome: Overall Survival (OS) of Patients Treated With Everolimus After Failure of First-line Sunitinib or Pazopanib Therapy up to 48 Months
Description: Overall survival (OS) was defined as the time from date of start of treatment to date of death due to any cause. If a patient was not known to have died, survival will be censored at the date of last contact.
Time Frame: 48 months
Population: Full Analysis Set (FAS) consisted of all patients who received at least one dose of everolimus.
Measure: Median (80% Confidence Interval); unit: months
Arm/Group | 1st Line SUN | 1st Line PAZ
Number analyzed (Participants) | 12 | 13
months | 14.8 [10.0 to NA] — upper CI could not be calculated due to too few events | 20.4 [13.6 to NA] — upper CI could not be calculated due to too few events

5. Secondary Outcome: Duration of Response (DOR) in Patients Treated With Everolimus After Failure of First-line Sunitinib or Pazopanib Therapy up to 48 Months
Description: The duration of overall response (DOR) was defined as the time from the first occurrence of a confirmed Complete Response (CR) or Partial Response (PR) (as per investigator assessment according to RECIST 1.1) until the date of the first documented disease progression or death due to underlying cancer. If a patient did not have an event or received any further anticancer therapy, duration of overall response was censored at the date of last adequate tumor assessment. Duration of response was displayed only for patients whose best overall response was CR or PR. As none of the patients showed any response (CR or PR), DOR could not be calculated
Time Frame: 48 months
Population: Duration of response was displayed only for patients whose best overall response was CR or PR. As none of the patients showed any response (CR or PR), DOR could not be calculated
Arm/Group | 1st Line SUN | 1st Line PAZ
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All adverse events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Groups:
- Everolimus All Patients: Everolimus - All Patients that failed 1st line SUN and 1st Line PAZ and was on Everolimus 10mg orally once daily
Arm/Group | 1st Line SUN | 1st Line PAZ | Everolimus All Patients
Serious Adverse Events (participants affected / at risk) | 6/16 | 8/13 | 14/29
Other Adverse Events (participants affected / at risk) | 15/16 | 13/13 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1st Line SUN (N=16) | 1st Line PAZ (N=13) | Everolimus All Patients (N=29)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 1 | 2
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 | 1 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 1
ENTEROCUTANEOUS FISTULA (Gastrointestinal disorders) | 1 | 0 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 1 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 0 | 1 | 1
VOMITING (Gastrointestinal disorders) | 1 | 0 | 1
ASTHENIA (General disorders) | 0 | 1 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 1 | 2
PYREXIA (General disorders) | 1 | 0 | 1
ABDOMINAL ABSCESS (Infections and infestations) | 1 | 0 | 1
ENDOCARDITIS (Infections and infestations) | 1 | 1 | 2
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 1 | 2
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1 | 1
DEMENTIA (Nervous system disorders) | 0 | 1 | 1
SYNCOPE (Nervous system disorders) | 0 | 1 | 1
POLYURIA (Renal and urinary disorders) | 1 | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1st Line SUN (N=16) | 1st Line PAZ (N=13) | Everolimus All Patients (N=29)
ANAEMIA (Blood and lymphatic system disorders) | 4 | 7 | 11
HAEMORRHAGIC DIATHESIS (Blood and lymphatic system disorders) | 0 | 1 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 0 | 1 | 1
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 1 | 1
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 1
EYELID OEDEMA (Eye disorders) | 1 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 0 | 2
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0 | 1
APHTHOUS ULCER (Gastrointestinal disorders) | 0 | 1 | 1
ASCITES (Gastrointestinal disorders) | 0 | 1 | 1
CONSTIPATION (Gastrointestinal disorders) | 1 | 1 | 2
DIARRHOEA (Gastrointestinal disorders) | 6 | 3 | 9
DRY MOUTH (Gastrointestinal disorders) | 1 | 0 | 1
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0 | 1
FLATULENCE (Gastrointestinal disorders) | 0 | 1 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1 | 1
LIP ULCERATION (Gastrointestinal disorders) | 0 | 1 | 1
NAUSEA (Gastrointestinal disorders) | 3 | 6 | 9
ORAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 1
ORAL PAIN (Gastrointestinal disorders) | 1 | 0 | 1
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 0 | 1 | 1
STOMATITIS (Gastrointestinal disorders) | 2 | 7 | 9
VOMITING (Gastrointestinal disorders) | 2 | 0 | 2
ASTHENIA (General disorders) | 1 | 0 | 1
CHILLS (General disorders) | 0 | 1 | 1
FACE OEDEMA (General disorders) | 1 | 1 | 2
FATIGUE (General disorders) | 5 | 7 | 12
FEELING COLD (General disorders) | 0 | 1 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 1 | 2
OEDEMA PERIPHERAL (General disorders) | 2 | 7 | 9
PYREXIA (General disorders) | 1 | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 1 | 1
CANDIDA INFECTION (Infections and infestations) | 1 | 0 | 1
CONJUNCTIVITIS (Infections and infestations) | 0 | 1 | 1
NASOPHARYNGITIS (Infections and infestations) | 1 | 1 | 2
PERITONITIS (Infections and infestations) | 1 | 0 | 1
PHARYNGITIS (Infections and infestations) | 0 | 1 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 1
RHINITIS (Infections and infestations) | 1 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 2 | 2 | 4
URINARY TRACT INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 | 0 | 3
BLOOD CHLORIDE DECREASED (Investigations) | 1 | 0 | 1
BLOOD CHLORIDE INCREASED (Investigations) | 1 | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 3 | 2 | 5
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 | 0 | 1
BLOOD PHOSPHORUS DECREASED (Investigations) | 1 | 0 | 1
CLOSTRIDIUM TEST POSITIVE (Investigations) | 1 | 0 | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 3 | 0 | 3
GLUCOSE URINE PRESENT (Investigations) | 1 | 0 | 1
HAEMATOCRIT DECREASED (Investigations) | 3 | 0 | 3
HIGH DENSITY LIPOPROTEIN DECREASED (Investigations) | 1 | 0 | 1
LOW DENSITY LIPOPROTEIN INCREASED (Investigations) | 1 | 0 | 1
NEUTROPHIL COUNT INCREASED (Investigations) | 1 | 0 | 1
PLATELET COUNT INCREASED (Investigations) | 1 | 0 | 1
RED BLOOD CELL COUNT DECREASED (Investigations) | 1 | 0 | 1
WEIGHT DECREASED (Investigations) | 2 | 1 | 3
CACHEXIA (Metabolism and nutrition disorders) | 0 | 1 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 5 | 5 | 10
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 2 | 2
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 3 | 1 | 4
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 2
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 3 | 0 | 3
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 1
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPOCHLORAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 2
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 2
PROTEIN DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 4 | 6
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
AGEUSIA (Nervous system disorders) | 1 | 0 | 1
DYSGEUSIA (Nervous system disorders) | 1 | 2 | 3
HEADACHE (Nervous system disorders) | 2 | 2 | 4
HYPOAESTHESIA (Nervous system disorders) | 1 | 0 | 1
HYPOGEUSIA (Nervous system disorders) | 0 | 1 | 1
NEURALGIA (Nervous system disorders) | 1 | 0 | 1
ORTHOSTATIC INTOLERANCE (Nervous system disorders) | 0 | 1 | 1
PARAESTHESIA (Nervous system disorders) | 1 | 0 | 1
POLYNEUROPATHY (Nervous system disorders) | 0 | 1 | 1
SYNCOPE (Nervous system disorders) | 0 | 1 | 1
TREMOR (Nervous system disorders) | 1 | 0 | 1
APATHY (Psychiatric disorders) | 1 | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 1 | 1
RESTLESSNESS (Psychiatric disorders) | 0 | 1 | 1
SLEEP DISORDER (Psychiatric disorders) | 1 | 0 | 1
INCONTINENCE (Renal and urinary disorders) | 1 | 0 | 1
NEPHROSCLEROSIS (Renal and urinary disorders) | 1 | 0 | 1
PROTEINURIA (Renal and urinary disorders) | 1 | 1 | 2
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 1
GENITAL TRACT INFLAMMATION (Reproductive system and breast disorders) | 1 | 0 | 1
PELVIC PAIN (Reproductive system and breast disorders) | 1 | 0 | 1
ALVEOLITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 | 5 | 11
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 7
DYSPNOEA AT REST (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 7
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
NASAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
PAINFUL RESPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 2 | 2
ECZEMA (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 3 | 5 | 8
RASH (Skin and subcutaneous tissue disorders) | 3 | 2 | 5
BLOOD PRESSURE FLUCTUATION (Vascular disorders) | 1 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 0 | 1
PERIPHERAL COLDNESS (Vascular disorders) | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.